CLINICAL TRIAL: NCT07030816
Title: Effects of Wearing a Lumbar Support Belt on Low-Back Pain, Physical Fatigue During Computer Use, and Work Performance: A Pilot Parallel-Group Randomised Controlled Trial
Brief Title: Lumbar Support Belt for Low-Back Pain in Office Workers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: General Incorporated Foundation Ryukyuseimeisaiseikai, Ryusei Hospital. (Other)
Responsible Party: Principal Investigator, Shinyu Kise, Principal Investigator , Institute for Tourism and Health, General Incorporated Foundation Ryukyuseimeisaiseikai, Ryusei Hospital.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202502
Record Dates: First submitted 2025-06-12; First posted 2025-06-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Low Back Pain (LBP); Chronic Low Back Pain; Non-specific Low Back Pain
Keywords: Lumbar support belt; Elastic lumbar belt; Office workers; Workplace intervention; Presenteeism; Fatigue; Randomised controlled trial
MeSH Terms: conditions — Low Back Pain; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lumbar Support Belt Group (Experimental): Participants wore a commercially available elastic lumbar support belt (Guardner Belt) sized according to waist circumference during working hours (≥ 8 hours/day) for 4 weeks.
  Interventions: Device: Guardner Belt
- Control Group (No Intervention): Participants continued their usual daily work routines without using any lumbar support belt.

INTERVENTIONS:
Device: Guardner Belt — The Guardner Belt is a commercially available elastic lumbar support belt designed to reduce low-back pain and improve posture. Participants wore the belt sized according to waist circumference for at least 8 hours per day during working hours for 4 weeks.
  Arms: Lumbar Support Belt Group

SUMMARY:
Background:

Low-back pain (LBP) is common among office workers and can reduce productivity and quality of life. Lumbar support belts are commonly used to manage LBP, but their effectiveness specifically for office workers remains uncertain.

Aim:

This study investigates whether wearing a commercially available lumbar support belt (Guardner Belt) can reduce low-back pain, decrease physical fatigue during computer work, and improve perceived work performance among office workers with chronic low-back pain.

Methods:

Thirty office workers with chronic nonspecific low-back pain were randomly assigned to either wear the lumbar support belt during work hours for four weeks or continue usual activities without the belt. Participants' pain, fatigue, and work performance were assessed before and after the intervention period.

DETAILED DESCRIPTION:
Study Design:

A single-centre, open-label, parallel-group randomised controlled trial conducted at a logistics company in Okinawa, Japan.

Participants:

Inclusion criteria: full-time office workers aged 20 to 65 years, chronic nonspecific low-back pain intensity ≥ 30 mm (100-mm visual analogue scale; VAS).

Exclusion criteria: prior lumbar surgery, ongoing pharmacologic treatment for low-back pain, anticipated changes in job duties during the trial period.

Interventions:

* Belt Group: Participants wore a commercially available elastic lumbar support belt (Guardner Belt) sized according to waist circumference. Participants were instructed to wear the belt for at least 8 hours daily during their working hours over a 4-week period.
* Control Group: Participants continued normal daily routines without any lumbar support belt.

Primary Outcome Measures:

Assessed at baseline and after 4 weeks of intervention:

* Low-back pain intensity: Measured using a 100-mm Visual Analogue Scale (VAS).
* Physical fatigue during computer work: Measured using a 100-mm VAS.
* Work performance: Measured using the Single-Item Presenteeism Question (SPQ), scored from 0% (no productivity) to 100% (full productivity).

Ethics:

Ethical approval was retrospectively granted by the Ryusei Hospital Institutional Review Board (Approval Number 202502). Written informed consent was obtained from all participants.

ELIGIBILITY:
Inclusion Criteria:

* • Full-time desk workers

  * Chronic nonspecific low-back pain (≥30 mm on a 100-mm visual analogue scale at baseline)
  * Age between 20 and 65 years

Exclusion Criteria:

* • Previous lumbar surgery

  * Currently receiving pharmacologic treatment for low-back pain
  * Planned job-duty changes during the study period

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Low Back Pain Intensity (VAS) | Baseline and Week 4
  Low back pain intensity assessed using a 100-mm Visual Analogue Scale (0 mm = no pain, 100 mm = worst imaginable pain).
Physical Fatigue During Computer Work (VAS) | Baseline and Week 4
  Physical fatigue during computer work assessed using a 100-mm Visual Analogue Scale (0 mm = no fatigue, 100 mm = extreme fatigue).
Self-rated Work Performance (SPQ) | Baseline and Week 4
  Self-rated work performance assessed using the Single-Item Presenteeism Question (0% = no productivity, 100% = full productivity).

CONTACTS AND LOCATIONS:
Locations (1):
- Ryusei Hospital, Naha, Okinawa, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Qaseem A, Wilt TJ, McLean RM, Forciea MA; Clinical Guidelines Committee of the American College of Physicians; Denberg TD, Barry MJ, Boyd C, Chow RD, Fitterman N, Harris RP, Humphrey LL, Vijan S. Noninvasive Treatments for Acute, Subacute, and Chronic Low Back Pain: A Clinical Practice Guideline From the American College of Physicians. Ann Intern Med. 2017 Apr 4;166(7):514-530. doi: 10.7326/M16-2367. Epub 2017 Feb 14. PMID 28192789